CLINICAL TRIAL: NCT02436980
Title: Effects of Midazolam or Tramadol Premedication on Early Cognitive Function in ERCP: a Randomized Controlled Double-Blind Study
Brief Title: Premedication for ERCP With Midazolam or Tramadol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Hulya ULUSOY, Assoc.Prof.Dr., Karadeniz Technical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 499
Record Dates: First submitted 2015-04-27; First posted 2015-05-07 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Chronic Disease
Keywords: premedication; ERCP; midazolam; tramadol; cognitive
MeSH Terms: conditions — Chronic Disease | interventions — Tramadol; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- tramadol (Active Comparator): 1mg/kg of tramadol drop (Contramal® drop, Abdi Ibrahim Ilaç San.,istanbul) was administered orally in 10 mL of cherry juice without particles in preparation room before intervention, Group T who were separated randomly to two premedication groups.
  Interventions: Drug: Tramadol
- midazolam (Active Comparator): 0.15 mg/kg of midazolam (Dormicum®, ampoule, Roche Products A.Ş., istanbul) was administered orally in 10 mL of cherry juice without particles in preparation room before intervention, to Group M who were separated randomly to two premedication groups.
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Tramadol — GROUP T
  Other Names: CONTRAMAL
  Arms: tramadol
Drug: Midazolam — GROUP M
  Other Names: DORMICUM
  Arms: midazolam

SUMMARY:
OBJECTIVE:Purpose of this study is to set forth the sedative efficacy and effects on early period cognitive functions of two premedication drugs used for ERCP (Endoscopic retrograde cholangiopancreatography) METHODS:This randomized and double blind study was performed with forty (18-70 of age) ASA I-III risk group patients for who elective ERCP was planned. Cognitive functions of patients were determined by mini-mental test (MMT). 0.5 mg/kg midazolam or 1mg/kg tramadol drop was administered orally before intervention to patients who were randomly divided into two premedication groups.

Vital signs,BIS (Bispectral index), mRSS (modified Ramsay Sedation scale), NRS (numeric rating scale ) was evaluated. If MMT (mini-mental test) was ≤ 23 at 60th minute it was considered as cognitive impairment. Recovery period, post-procedure state of cognitive function at 60th minute were recorded.

DETAILED DESCRIPTION:
The Outcome Measures are number of Participants with Adverse Events, and the incidence of Postoperative cognitive dysfunction assessed by MMT (mini-mental test) in first 60 minutes.

ELIGIBILITY:
Inclusion Criteria:

* This study was conducted in the Endoscopy Department for forty (18-70 years old) outpatients in ASA I-III risk group were randomized and double blind planned for elective ERCP.

Exclusion Criteria:

* American Society of Anesthesiologist (ASA) class greater than 3,
* morbid obesity,
* major organ dysfunction (respiratory, renal and hepatic),
* history of drug addiction,
* known hypersensitivity for tramadol, midazolam and remifentanil,
* mini-mental test (MMT) ≤ 23 or
* refusal of the patient.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-01; Primary Completion 2009-09 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
The early cognitive functions after ERCP | Postprocedure in the first 60 minutes
  The early cognitive functions after ERCP assessed by mini-mental test (MMT)

SECONDARY OUTCOMES:
Number of Participants with Adverse Events | Postprocedure in first 60 minutes
  With any side effects

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Arslan, Prof.Dr., Study Chair — Gastroenterology Department